CLINICAL TRIAL: NCT06449326
Title: Multimodal Image Analysis and Guidance of Neuromodulation for Trauma-Related Symptoms
Acronym: MAGNETS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: New Mexico VA Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-451
Record Dates: First submitted 2024-05-06; First posted 2024-06-10 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, parallel-design, sham-controlled clinical trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active iTBS (Active Comparator): Participants in this arm will undergo 50 sessions of active accelerated (10x/day, five days) image-guided iTBS.
  Interventions: Device: Active Intermittent theta burst stimulation
- Sham iTBS (Sham Comparator): Participants in this arm will undergo 50 sessions of sham accelerated (10x/day, five days) image-guided iTBS.
  Interventions: Device: Sham Intermittent theta burst stimulation

INTERVENTIONS:
Device: Active Intermittent theta burst stimulation — Intermittent theta burst stimulation (iTBS) is an efficient form of transcranial magnetic stimulation that allows up to 10x more pulses to be delivered in a given timeframe compared to conventional stimulation patterns.
  Arms: Active iTBS
Device: Sham Intermittent theta burst stimulation — Intermittent theta burst stimulation (iTBS) is an efficient form of transcranial magnetic stimulation that allows up to 10x more pulses to be delivered in a given timeframe compared to conventional stimulation patterns.
  Arms: Sham iTBS

SUMMARY:
MAGNETS is a prospective, randomized, parallel-design, sham-controlled clinical trial of accelerated, functional magnetic resonance imaging (fMRI)-guided intermittent theta burst stimulation (iTBS) to the right dorsolateral prefrontal cortex (dlPFC) for chronic symptoms of posttraumatic stress disorder (PTSD) in a comorbid Veteran population.

DETAILED DESCRIPTION:
In MAGNETS, sixty-four participants will be recruited from the NMVAHCS PTSD programs, Polytrauma services, and outpatient mental health clinics. At study entry (Visit #1), participants will undergo baseline demographic, behavioral, and cognitive assessment, and fMRI and diffusion tensor imaging (DTI). The data analysis team will then determine the image-based target in the right hemisphere. Participants will be randomized to either the active (n=32) or sham (n=32) group and undergo 50 sessions of iTBS (10x/day, five days). At end of treatment (Visit #2), they will repeat all baseline tests, including fMRI. One-, three- and six-month symptom levels will be obtained through phone visits (Visits #3-5) to establish longevity and stability of benefit. Repeated measures analyses will be performed on behavioral and connectivity variables, with clinical (age, duration, head injury history) and imaging (white matter fiber counts) features as covariates.

ELIGIBILITY:
Inclusion Criteria:

* Veterans will be enrolled in this study if they:

  1. are aged 18-80;
  2. have a documented diagnosis of PTSD with evidence of ongoing symptoms as demonstrated by score of "31" or higher on the PCL-5, a measure of posttraumatic stress symptoms;
  3. are fluent in English (as the neuropsychological testing tools used are only available in English) and
  4. have been on stable doses of psychotropic medications for the past month.

Exclusion Criteria:

* Veterans will be excluded from participation in this study if there is:

  1. a prior history of other neurological disease beyond mild TBI, as determined by VA/DoD criteria for TBI severity;
  2. any history of seizures beyond immediate posttraumatic seizure or childhood febrile seizure, so as to reduce risk of exacerbation of epilepsy or other neurological symptoms;
  3. history of a psychotic disorder, such as schizophrenia or bipolar disorder, so as to reduce risk of psychiatric decompensation;
  4. active substance/alcohol dependence without ongoing treatment, to reduce confounding effects on diagnosis and brain imaging;
  5. presence of any implanted electrical device (e.g., pacemaker), to reduce risk of device malfunction from rTMS;
  6. recent medical hospitalization (within four weeks), to reduce risk of medical decompensation during the study;
  7. any condition that would prevent the subject from completing the protocol;
  8. appointment of a legal representative or inability to provide informed consent, to avoid coercion of a vulnerable population;
  9. any ongoing litigation related to PTSD, TBI, disability determination, or service connection, to prevent interference with legal proceedings;
  10. any contraindication to MRI;
  11. pregnant women, so as to prevent complications;
  12. membership in an identified vulnerable population, including minors and prisoners, so as to prevent coercion;
  13. Cognitively impaired adults who lack capacity to consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
CAPS-5 | Immediate post-treatment visit
  Clinician Administered PTSD Scale-DSM 5 (range 0-80; higher scores = more symptoms)

SECONDARY OUTCOMES:
PCL-5 | Immediate post-treatment visit, 1 month, 3 months, 6 months
  PTSD Checklist-DSM 5 (range 0-80; higher scores = more symptoms)
PHQ-9 | Immediate post-treatment visit, 1 month, 3 months, 6 months
  Patient Health Questionnaire-9 (range 0-27; higher scores = more symptoms)
GAD-7 | Immediate post-treatment visit, 1 month, 3 months, 6 months
  Generalized Anxiety Disorder-7 (range 0-21; higher scores = more symptoms)
NSI | Immediate post-treatment visit, 1 month, 3 months, 6 months
  Neurobehavioral Symptom Inventory (range 0-88; higher scores = more symptoms)
DSM-XC (range 0-92; higher scores = more symptoms) | Immediate post-treatment visit, 1 month, 3 months, 6 months
  Diagnostic and Statistical Manual Cross-Cutting Assessment
WHODAS | Immediate post-treatment visit, 1 month, 3 months, 6 months
  World Health Organization Disability Assessment Schedule (range 0-100; higher scores = more disability)
PGIC | Immediate post-treatment visit, 1 month, 3 months, 6 months
  Patient Global Impression of Change (range 0-7; higher scores = more positive change)

OTHER OUTCOMES:
AIM | Immediate post-treatment visit
  Acceptability of Intervention Measure, a four-item measure of the acceptability of an intervention. It has five questions, scored on a 5-point Likert scale, from "completely disagree" to "completely agree"
fMRI Connectivity | Immediate post-treatment visit
  Connectivity between the dlPFC and vmPFC (range -1.0 to 1.0; higher scores indicate greater degree of positive correlation

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UNM Center for Psychiatric Research, Albuquerque, New Mexico
  - New Mexico VA Health Care System, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: Undecided